CLINICAL TRIAL: NCT03803215
Title: Theophylline in Patients With Unexplained Syncope and Low Adenosine. Study Verified by ICM, Controlled by Propensity-score Matching
Brief Title: Theophylline for Low Adenosine Syncope
Acronym: THEO-USA
Status: Completed | Type: Observational
Sponsor: Centro Prevenzione Malattie Cardiovascolari N. e V. Corbella (Other)
Collaborators: Gruppo Italiano Multidisciplinare per lo Studio della Sincope (Other)
Responsible Party: Sponsor
Other Study IDs: CPM 30102018
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-01

CONDITIONS: Syncope
Keywords: theophylline; asystole; implantable loop recorder
MeSH Terms: conditions — Syncope; Heart Arrest | interventions — Theophylline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Theophylline group: Patients who have electrocardiographic documentation of asystolic syncope will be treated with oral theophylline at tailored dosage
  Interventions: Drug: Theophylline
- Control untreated group: A propensity-score matched control group is generated from the large database of patients who had received an implantable loop recorder

INTERVENTIONS:
Drug: Theophylline — Oral theophylline initially 600 mg bid and then titrated at the maximum tolerated dose
  Groups: Theophylline group

SUMMARY:
The study aims at assessing that theophylline is effective in patients with no prodromes, normal heart and with low values of plasmatic adenosine compared with a propensity-score matched untreated control population who have received an implantable cardiac monitor (ICM) for diagnosis of unexplained or atypical reflex syncope.

DETAILED DESCRIPTION:
Theophylline has been used for 3 decades in ordinary medical practice to tentatively prevent syncopal recurrences in patients affected by neurally-mediated syncope. Observational studies report a recurrence rate with this drug ranging between 12% and 22%. Theophylline was much more effective in selected patients with syncope without prodromes and normal heart who had ECG documentation of long pauses at the time of syncopal attack and low values of baseline plasmatic adenosine. Since theophylline is a non-selective antagonist of purinergic receptors, it has been hypothesized that purinergic receptors are involved in the mechanism of syncope in such patients. Conversely, theophylline was suspected to be ineffective (or less effective) in patients affected by other forms of neurally-mediated syncope.

The present study aims at assessing that theophylline is effective in patients with no prodromes, normal heart and with low values of plasmatic adenosine compared with a propensity-score matched untreated control population.

This will be a multicenter, non interventional study, verified by ICM, with 2 predefined subgroups:

Subgroup #1

* Low adenosine group: Patients with Low Adenosine values (<0.40 μmol/L)
* Normal/high adenosine (≥0.40 μmol/L) group: any other patient Subgroup #2
* Patients with no prodromes or very short prodromes (≤5 sec), normal heart and normal ECG (No prodrome group)
* Any other form of atypical neurally-mediated syncope with prodromes >5 sec. Remote or in-hospital periodic follow-up will be done according to centre's clinical practice for ICM monitoring.

Patients will be followed up until the first primary endpoint event with a maximum follow-up of 24 months since start of theophylline treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female gender with age >18 years
2. Unexplained syncope without prodrome or neurally-mediated syncope with atypical prodrome, with normal heart and normal ECG
3. Two syncopes /last year or 3 syncopes /last 2 years before start of theophylline treatment
4. Having received an ICM according to conventional guideline-based indications
5. Being treated with oral theophylline therapy, while been waiting for ICM diagnosis
6. Having signed a written informed consent to the study participation and to the treatment of personal data

Exclusion Criteria:

1. Typical vaso-vagal syncope with long prodromes and situational syncope
2. Any other form of syncope/T-LOC different from reflex syncope
3. Pregnant or breast-feeding patients -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received an implantable cardiac monitor (ICM) for diagnosis of unexplained or atypical reflex syncope
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Asystolic syncope | 24 months
  Number of patients. The primary objective aims to test the hypothesis that theophylline is able to reduce asystolic events in the Low-Adenosine subgroup compared with the propensity-score matched control group

SECONDARY OUTCOMES:
Time to first syncope recurrence | 24 months
  Months from enrolment to the first recurrence of syncope
Asystolic syncope in the subgroup with low adenosine plasmatic values | 24 months
  Number of patients with asystolic syncope during follow-up
Asystolic syncope in patients without prodrome, normal heart and normal ECG | 24 months
  Number of patients with asystolic syncope during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, MD, Principal Investigator — Department of Cardiology, Ospedali del Tigullio
Locations (1):
- Department of Cardiology, Ospedali del Tigullio, Lavagna, Italy

REFERENCES:
- [Derived] Brignole M, Iori M, Strano S, Tomaino M, Rivasi G, Ungar A, Carretta D, Solari D, Napoli P, Deharo JC, Guieu R. Theophylline in patients with syncope without prodrome, normal heart, and normal electrocardiogram: a propensity-score matched study verified by implantable cardiac monitor. Europace. 2022 Jul 21;24(7):1164-1170. doi: 10.1093/europace/euab300. PMID 34849728